CLINICAL TRIAL: NCT02638246
Title: Incentives for Internet-based Glucose Testing in Adolescent Type 1 Diabetes
Brief Title: Incentives for Internet-based Adherence to SMBG for Teens With T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rowan University (Other)
Collaborators: National Development and Research Institutes, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21HD061683-02 (NIH)
Record Dates: First submitted 2015-12-17; First posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Contingent Versus Noncontingent Incentives
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contingent (Experimental): Participants in this group received incentives contingent on meeting pre-specified daily blood-glucose testing adherence goals.
  Interventions: Behavioral: Internet-delivered, Incentive-based intervention + Motivational Interviewing
- Noncontingent (Active Comparator): Participants in this group received incentives independent of meeting pre-specified daily blood glucose testing adherence goals.
  Interventions: Behavioral: Internet-delivered, non-contingent incentives + Motivational Interviewing

INTERVENTIONS:
Behavioral: Internet-delivered, Incentive-based intervention + Motivational Interviewing — Blood glucose monitoring was verified by videos uploaded to a secure server. Participants in the experimental group received incentives for adherence whereas participants in the control group received adherence independent of adherence.
  Arms: Contingent
Behavioral: Internet-delivered, non-contingent incentives + Motivational Interviewing
  Arms: Noncontingent

SUMMARY:
Self-management of diabetes can result in long-term benefits, such as delaying or preventing the development of a number of unnecessary health complications, and can even reduce the chances of premature death. Because adherence to diabetes self-management often declines during adolescence, it is critically important to develop interventions that increase adherence of diabetes self-management skills in this population.

DETAILED DESCRIPTION:
Intensive glycemic control among diabetics decreases the risk of both the development and progression of a number of medical complications associated with diabetes. Self-monitoring blood glucose is a critical component of diabetes self-management and is correlated with improvements in glycemic control. Nevertheless, adherence to blood glucose monitoring is generally poor, particularly among youth, with one study reporting that only ~ 25% of adolescents adhered to the recommended frequency of blood glucose testing.

The current study will use a powerful, scientifically-based behavioral intervention - contingency management (CM) to increase self-monitoring of blood glucose and improve glycemic control among adolescents with Type 1 diabetes. CM involves giving incentives for objective evidence of a target behavior and has been shown to have a robust and reliable impact in promoting behavior change. Our previous research used the Internet to objectively monitor smoking and reinforce smoking cessation (via video recorded carbon monoxide submissions), which resulted in robust increases in smoking abstinence. The current proposal extends this effective Internet-based CM intervention to address the significant health issue of non-adherence to blood glucose testing and glycemic control among youth. Two groups of non-adherent adolescents will be recruited. One group will earn incentives over the Internet for submitting webcam recorded videos that show them testing their blood glucose. A different group will be given standard care recommendations for blood glucose testing and management and will be encouraged to submit glucose monitoring videos, but incentives will not be delivered contingent on submissions (instead, they will earn monetary incentives independent of video submissions, but in an overall amount that matches the earnings of a participant in the other group). The purpose of the study is to evaluate the feasibility, convenience, and efficacy of using Internet-based CM to increase blood glucose monitoring in adolescent Type 1 diabetics.

Combining the accessibility of the Internet with a powerful, evidence-based behavioral intervention can have profound effects on adherence to diabetes self-management in this important population. Improving adherence to diabetes management in adolescents is a significant public health issue - serious medical complications, such as heart disease and nerve damage, that would develop with poor glycemic control can be avoided. Importantly, the current study offers a scientifically-based behavioral intervention that could be applied to a range of populations and behavior relevant to adherence with diabetes regimens (e.g., adults, medication adherence, carbohydrate counting, insulin dose adjustment, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 1 diabetes for at least one year
* Self-reported self-monitoring blood glucose less than four times per day
* Lived in a home with Internet access
* No travel plans within 2 months of enrolling in the study
* Read and spoke English

Exclusion Criteria:

* Diagnosis other Type 1 diabetes within one year of screening
* Not attending regular clinic appointment within 3 months of screening

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Daily frequency of self-monitoring blood glucose | 45 days
Percentage of days conducted at least 4 tests per day. | 45 days

SECONDARY OUTCOMES:
Acceptability of the intervention | 45 days
  This was measured using a Treatment Acceptability Questionnaire
Feasibility | 45 days
  Feasibility was based on willingness to participate (recruitment), adherence with the video submission protocol, and attrition

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Raiff, PhD, Principal Investigator — Rowan University

IPD SHARING:
Plan to Share IPD: No
Only upon request